CLINICAL TRIAL: NCT01852851
Title: Employment and Arthritis: Making it Work: A Randomized Controlled Trial Evaluating an On-line Program to Help People With Inflammatory Arthritis Remain Employed
Brief Title: Employment and Arthritis: Making it Work
Acronym: MIW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); University of Toronto (Other); University of Calgary (Other); Simon Fraser University (Other)
Responsible Party: Principal Investigator, Diane Lacaille, Principal Investigator, University of British Columbia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: H11-03527
Record Dates: First submitted 2012-04-13; First posted 2013-05-14 (Estimated); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Rheumatoid Arthritis; Ankylosing Spondylitis; Lupus Erythematosus, Systemic; Psoriatic Arthritis; Other Connective Tissue Diseases; Spondylarthropathy
MeSH Terms: conditions — Arthritis, Rheumatoid; Spondylitis, Ankylosing; Lupus Erythematosus, Systemic; Arthritis, Psoriatic; Spondylarthropathies | interventions — Employment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention Group (Active Comparator): The intervention group will participate in the on-line eLearning program, an ergonomic assessment by an Occupational Therapist and job retention vocational counselling by a Vocational Rehabilitation Counsellor
  Interventions: Behavioral: Employment and Arthritis: Making it Work
- Control Group (No Intervention): The control group will receive "usual care" and receive printed educational materials about work and arthritis.

INTERVENTIONS:
Behavioral: Employment and Arthritis: Making it Work — A ten week on-line eLearning program designed to help people with inflammatory arthritis stay employed. The program consists of 1) 5 interactive web-based eLearning modules that participants will complete individually in between the weekly group sessions, 2) 5 weekly group sessions conducted as virtual real-time web-based group meetings led by a trained facilitator, 3) asynchronous communications such as a message board to facilitate additional interactions among participants, 4) consultations with an occupational therapist (in-person)for an ergonomic assessment, and a vocational rehabilitation counsellor (on-line consultation using web technology) for job retention vocational counselling.
  Arms: Intervention Group

SUMMARY:
The investigators plan to conduct a randomized controlled trial to evaluate the effectiveness and the cost effectiveness of an on-line eLearning program (entitled Employment and Arthritis: Making it Work) designed to help people with inflammatory arthritis stay employed. The program also includes assessments with 1) an occupational therapist, and 2) a vocational rehabilitation counsellor at the end of the program to help participants identify and obtain necessary changes at work. People from three provinces will be recruited from collaborators' patient and program recipient lists. The study group will receive the program intervention and the control group will receive "usual care" and printed educational material. All participants will be followed for five years. The effectiveness of the program at improving at work productivity and reducing work cessation will be evaluated compared to a control group receiving printed material on employment and arthritis.

ELIGIBILITY:
Inclusion Criteria:

* Between ages 18 and 59 years
* Able to read and write English
* Have inflammatory arthritis confirmed by a rheumatologist (Rheumatoid Arthritis, Ankylosing Spondylitis, Lupus Erythematosus, Systemic, Psoriatic Arthritis, Other Connective Tissue Diseases and Spondylarthropathy)
* Have access to a computer, a web-cam, a headset and a printer, or willingness to purchase these items
* Are willing to travel to Vancouver, Kelowna, Victoria, Prince Rupert, Prince George, Cranbrook or Kamloops, Calgary, Toronto, Newmarket or Brampton for one visit with an occupational therapist

Exclusion Criteria:

* Individuals who are not working
* Individuals on sick leave, short term or long term work disability
* Students
* People performing unpaid work such as volunteer work or taking care of family
* People planning to retire in the next six years
* Individuals unable to provide informed consent
* Individuals living outside of British Columbia, Alberta, Ontario

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 528 (Actual)
Dates: Start 2013-06; Primary Completion 2022-10 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Efficacy analysis of at work productivity | 2 years post intervention
  Primary outcome for efficacy analysis of at-work productivity will be measured using the Work Instability Scale (WIS)
Efficacy analysis of work cessation | Over 5 years of follow up
  Primary outcome for efficacy analysis of work cessation is time to complete work cessation, defined as complete cessation of work due to any reason, for at least six months.
Cost effectiveness analysis of at work productivity | 2 years post intervention
  Primary outcome for cost effectiveness analysis of at work productivity will be measured using the Work Productivity and Activity Impairment (WPAI)

SECONDARY OUTCOMES:
Temporary work cessation | Up to 5 years
  Time to temporary cessation of work for any reason (E.g. sick leave or temporary work disability and short periods of unemployment) for more than 2 months but less than 6 months
Occasional work absence | Up to 5 years
  Number of days missed from work per year, measured by self report
Reduction in usual amount of time worked | Up to 5 years
  Reduction in hours per week worked per year, measured by self report
Changes in employment risk factors | Up to 5 years
  Changes from baseline in job satisfaction, self-efficacy at work, work-related risk factors for work disability (physical demand, job autonomy, difficulty commuting, self-employment and support from co-workers, employers and family), job accommodations and job type, measured by self report
At-work productivity | Up to 5 years
  Evaluating maintenance of effect on at work productivity over 5 years using the Work Instability Scale (WIS)
At work productivity | Up to 5 years
  Evaluating maintenance of effect on at work productivity over 5 years using the Work Productivity and Activity Impairment (WPAI)
At work productivity | Up to 5 years
  New scale being developed and validated to measure at work productivity. Based on a combination of Workplace Activity Limitations Scale (WALS) and Work Limitations Questionnaire (WLQ).
Cost utility analysis of at work productivity | 2 years post intervention
  Outcome for cost utility analysis of at work productivity will be quality adjusted life year (QALY) measured using EQ-5D.
Cost utility analysis of at work productivity | 2 years post intervention
  Outcome for cost utility analysis of at work productivity will be quality adjusted life year (QALY) measured using SF-6D.

CONTACTS AND LOCATIONS:
Overall Officials: Diane Lacaille, MD, FRCPC, MHSc, Principal Investigator — University of British Columbia and Arthritis Research Centre
Locations (1):
- Arthritis Research Centre, Richmond, British Columbia, Canada

REFERENCES:
- [Derived] Carruthers EC, Rogers P, Backman CL, Goldsmith CH, Gignac MA, Marra C, Village J, Li LC, Esdaile JM, Lacaille D. "Employment and arthritis: making it work" a randomized controlled trial evaluating an online program to help people with inflammatory arthritis maintain employment (study protocol). BMC Med Inform Decis Mak. 2014 Jul 21;14:59. doi: 10.1186/1472-6947-14-59. PMID 25043631